CLINICAL TRIAL: NCT03694834
Title: Window of Opportunity Pilot Study of Pembrolizumab in Obesity-driven Endometrial Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC 1739
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Cancer; Uterine Cancer
Keywords: Endometrial Cancer; Uterus; Endometrioid
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — pembrolizumab; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm - Pembrolizumab (Experimental): Single dose of Pembrolizumab 200mg IV administered prior to hysterectomy and surgical staging.
  Interventions: Drug: Pembrolizumab; Procedure: Hysterectomy

INTERVENTIONS:
Drug: Pembrolizumab — A single dose of Pembrolizumab (200 mg) will be administered IV over 30 min (-5 /+10 min) approximately 3 weeks prior to the scheduled hysterectomy.
  Pembrolizumab (200 mg) will be administered IV over 30 min (-5/+10 min) every three weeks in combination with paclitaxel and carboplatin as adjuvant therapy over 6 cycles. Pembrolizumab should be given on D1 of each cycle after the infusion of cytotoxics.
  Other Names: Keytruda
Procedure: Hysterectomy — Hysterectomy/Surgical Staging per institutional standard of care.

SUMMARY:
Programmed cell death 1 (PD-1) inhibitor treatment may benefit patients with endometrial cancer (EC) based on the following observations: 1) an overwhelming presence of PD-1 in ECs; 2) the well-known effect of obesity which activates pro-inflammatory white blood cells and promotes the development of ECs; and 3) the high prevalence of a specific gene pattern (ie, microsatellite instability hypermutated [MSI high]) among ECs that may be particularly sensitive to this class of drugs. To identify potential biomarkers of response to PD-1 inhibitors in EC, we will conduct a window of opportunity study of pembrolizumab in 20 patients with clinical stage 1, grade 3 EC, encompassing endometrioid, serous and clear cell histologies. Eligible patients will undergo a research biopsy for collection of fresh tissue at the time of enrollment, in addition to the routinely performed endometrial biopsy that led to the diagnosis of their cancer. Patients will receive a single dose of pembrolizumab (200 mg IV) prior to undergoing their scheduled hysterectomy with surgical staging three weeks later. As per standard of care, adjuvant chemotherapy with paclitaxel and carboplatin will be recommended after hysterectomy/surgical staging for women with endometrioid tumors and stage III disease or women with serous/clear cell tumors at all stages of disease. However, in this study pembrolizumab will be added to adjuvant paclitaxel and carboplatin for EC. Pre-treatment endometrial biopsy specimens (fresh frozen tissue and formalin-fixed paraffin embedded (FFPE)) and a post-treatment hysterectomy specimen (fresh frozen tissue and FFPE) will be collected for translational studies. Blood, fecal and vaginal samples will be collected pre-treatment, at the time of surgery and following 3 cycles of adjuvant pembrolizumab/paclitaxel/carboplatin treatment.

DETAILED DESCRIPTION:
The primary objective of the trial is to measure the change in number and phenotype of tumor-infiltrating lymphocytes, including delineation of effector and regulatory T cells, before and after one cycle of pembrolizumab treatment. Other correlative secondary objectives include investigation of associations among pre-treatment TIL numbers, clonality of TILs and change in number and phenotype of TILs with samples collected after pembrolizumab treatment between MSI and DNA polymerase (POLE) ultramutated ECs versus MSI low/stable ECs versus copy number high (CNH) ECs, among others. To assess the complex interplay between obesity, molecular subtype, the microbiome and immune regulation, gut, vaginal and uterine microbiota profiles will be characterized and potential associations with body mass index (BMI), pre-treatment TIL numbers, clonality of TILs and change in the number and phenotype of TILs will be investigated. Secondary clinical objectives include (1) of the pathologic response rate after one cycle of pembrolizumab following hysterectomy and surgical staging in stage I/II, serous/clear cell EC and stage III, G3 (serous, clear cell or endometrioid histologies) EC and (2) characterization of the toxicity profile of pembrolizumab pre-hysterectomy and in combination with paclitaxel and carboplatin as adjuvant therapy for EC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Female Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 1 (See Appendix 11.4).
* Diagnosis of advanced stage and histologically confirmed endometrioid, serous, clear cell, carcinosarcoma (including mixed) cancer of the uterus in which neoadjuvant chemotherapy is planned.
* Has received no prior therapy for uterine cancer, including hysterectomy
* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 72 hours prior to initiating study treatment.
* Have an available endometrial biopsy for correlative studies and willing to undergo a research biopsy prior to initiating study treatment. The research biopsy procedure must be deemed medically safe by the investigator.
* Subjects is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.

Exclusion Criteria:

* Active infection requiring systemic therapy.
* Pregnant or breastfeeding
* Has received a live vaccine within 30 days prior to the first dose of study drug.

Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Subject is receiving prohibited medications or treatments that cannot be discontinued/replaced by an alternative therapy.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen; HBsAg reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has a history of symptomatic congestive heart failure (e.g. congestive heart failure defined as New York Heart Association (NYHA) Class III or IV functional status), unstable angina pectoris or cardiac arrhythmia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Change in the number of Tumor Infiltrating Lymphocytes | 3 weeks
  Change in number of tumor-infiltrating lymphocytes in response to single dose of pembrolizumab will be determined by performing histopathologic analysis of H&E-stained tumor sections collected at baseline and at the time of surgery.

SECONDARY OUTCOMES:
Number of patients who experience Adverse Events after one dose of Pembrolizumab | 3 weeks
  The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Change in number of Tumor Infiltrating Lymphocytes by endometrial cancer sub-types | 3 weeks
  Count and compare associations of (1) pre-treatment Tumor Infiltrating Lymphocyte (TIL) numbers (2) clonality of TILs and (3) change in number and phenotype of TILs with pembrolizumab treatment between Microsatellite Instability (MSI) and DNA Polymerase ε Endometrial Cancers (EC) versus MSI low/stable ECs versus Copy Number High ECs.
Correlation of Programmed Cell Death-1 (PD-1) Expression with TILs | 3 weeks
  Compare possible associations of PD-1, Programmed Death Ligand 1 (PD-L1) and Programmed Death Ligand 2 (PD-L2) messenger Ribonucleic Acid (mRNA) expression with (1) pre-treatment TIL numbers (2) clonality of TILs and (3) change in number and phenotype of TILs.
Correlation of Immune and Obesity/Inflammation EC Signatures with TILs | 3 weeks
  Compare possible associations of immune and obesity/inflammation EC signatures with (1) Body Mass Index (BMI) (2) pre-treatment TIL numbers (3) clonality of TILs and (4) change in number and phenotype of TILs.
Correlation of Microbiota Profiles with TILs | 3 weeks
  Compare possible associations of gut, vaginal and uterine microbiota profiles with (1) BMI (2) pre-treatment TIL numbers (3) clonality of TILs and (4) change in number and phenotype of TILs.
Overall Response Rate of Pembrolizumab with Paclitaxel and Carboplatin | 3 weeks
  Calculate the overall response rate of pembrolizumab in combination with paclitaxel and carboplatin following hysterectomy and surgical staging in (1) stage I/II, serous/clear cell EC and (2) stage III, Grade 3 (serous, clear cell or endometrioid histologies) EC.
  Response is measured as:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis <10mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bae-Jump, MD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials